CLINICAL TRIAL: NCT05047029
Title: Multiparametric Magnetic Resonance Imaging in Patients With Liver Cirrhosis for Evaluation of Myocardial Fibrosis and Inflammation in Cirrhotic Cardiomyopathy
Brief Title: Myocardial Fibrosis and Inflammation in Liver Cirrhosis
Status: Completed | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Julian Alexander Luetkens, Prinicipal Investigator, Senior Physician, University Hospital, Bonn
Other Study IDs: 282/18_1
Record Dates: First submitted 2021-09-08; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Cirrhosis, Liver; Cardiomyopathies; Portal Hypertension
MeSH Terms: conditions — Liver Cirrhosis; Cardiomyopathies; Hypertension, Portal | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with cirrhosis: Patients with cirrhosis and transjugular intrahepatic portosystemic shunt implantation.
  Interventions: Procedure: Transjugular intrahepatic portosystemic shunt implantation; Diagnostic Test: Magnetic resonance imaging

INTERVENTIONS:
Procedure: Transjugular intrahepatic portosystemic shunt implantation — Transjugular intrahepatic portosystemic shunt is an artificial channel within the liver that establishes communication between the inflow portal vein and the outflow hepatic vein. It is used to treat portal hypertension (e.g., in liver cirrhosis)
Diagnostic Test: Magnetic resonance imaging — Multiparametric cardiac and hepatic magnetic resonance imaging

SUMMARY:
The aim of this clinical prospective study is to assess structural and functional myocardial changes in patients with liver cirrhosis after implantation of transjugular intrahepatic portosystemic shunt (TIPS).

ELIGIBILITY:
Inclusion criteria:

* liver cirrhosis with evaluation of TIPS implantation
* patients who are 18 years of age or older

Exclusion criteria:

* underlying cardiac disease, e.g. known myocardial infarction, previous myocarditis, congenital heart disease, cardiomyopathies of other causes known underlying disease witt potential cardiac involvement, e.g. storage disease (e.g. hemochromatosis, Fabry disease), inflammatory (e.g. sarcoidosis), endocrinological (e.g. diabetes mellitus, hyper-/hypothyroidism), autoimmune (e.g. systemic lupus erythematosus, dermatomyositis, rheumatoid arthritis), therapeutic (chemotherapy).
* patients with contraindication for contrast-enhanced MRI
* pregnant and breastfeeding women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Primary care clinic (Department of Internal Medicine I, University Hospital Bonn, Germany)
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
Myocardial T1 relaxation time | Change after 1 year of transjugular intrahepatic portosystemic shunt insertion.
  T1 relaxation times will be obtained to asses acute myocardial injury and fibrosis. T1 maps will be analyzed using a segmental approach by region of interest analysis. T1 relaxation times are given in [ms].

SECONDARY OUTCOMES:
Myocardial T2 relaxation time | Change after 1 year of transjugular intrahepatic portosystemic shunt insertion.
  T2 relaxation times will be obtained to asses myocardial edema. T2 maps will be analyzed using a segmental approach by region of interest analysis. T2 relaxation times are given in [ms].
Myocardial ECV | Change after 1 year of transjugular intrahepatic portosystemic shunt insertion.
  Myocardial extracellular volume will be obtained to asses extracellular space/myocardial fibrosis. ECV values will be calculated using a segmental approach by region of interest analysis of native and contrast-enhanced T1 relaxation maps. ECV values are given in [%].

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Hospital Bonn, Clinic for Diagnostic and Interventional Radiology, Bonn, North Rhine-Westphalia
  - University Hospital Bonn, Medical Clinic and Polyclinic I, Bonn, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Isaak A, Praktiknjo M, Jansen C, Faron A, Sprinkart AM, Pieper CC, Chang J, Fimmers R, Meyer C, Dabir D, Thomas D, Trebicka J, Attenberger U, Kuetting D, Luetkens JA. Myocardial Fibrosis and Inflammation in Liver Cirrhosis: MRI Study of the Liver-Heart Axis. Radiology. 2020 Oct;297(1):51-61. doi: 10.1148/radiol.2020201057. Epub 2020 Aug 18. PMID 32808886